CLINICAL TRIAL: NCT00912782
Title: Impact of Vitamin D on Arteriovenous Fistulae Maturation Among ESRD Patients
Brief Title: Vitamin D and Arteriovenous Fistulae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Monnie Wasse MD, MPH, FASN, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00014859
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: End-stage Renal Disease
Keywords: ESRD; Vitamin D; Arteriovenous Fistulae; Dialysis Vascular Access
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo one time per week for 3 weeks
  Interventions: Drug: Placebo
- Cholecalciferol (Experimental): Vitamin D 200,000 IU per week for 3 weeks
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 200,000 IU once a week for 3 weeks
  Arms: Cholecalciferol
Drug: Placebo — Placebo one time per week for 3 weeks
  Arms: Placebo

SUMMARY:
Patients requiring hemodialysis following kidney failure need a form of dialysis vascular access in order to undergo the dialysis procedure. Dialysis vascular access dysfunction is an enormous clinical problem. While the best form of vascular access is the arteriovenous fistula (AVF), its primary problem is early, aggressive cellular ingrowth that leads to poor maturation of the vessel, preventing its use for dialysis. Strategies to prevent AVF failure are needed.

Vitamin D is a hormone present in all human bodies and is important for good bone formation and immune function. There is new information that links vitamin D to the function of our veins and arteries, which are used in the creation of an arteriovenous fistulae. Our bodies can make vitamin D and can also get vitamin D from our diet. However, a majority of patients with chronic kidney disease and end-stage renal disease (ESRD) have low vitamin D levels (vitamin D deficiency). There are several benefits to correcting low vitamin D levels, however, it is not know whether correcting low vitamin D in the body will lead to better function of the vein and artery used for arteriovenous fistulae creation. The main goal of this pilot study is to examine the role of vitamin D supplementation on AVF maturation and useability for dialysis. Study results will be used to develop larger studies to examine the specific effect that vitamin D supplementation has on the vessels used for AVF creation and whether vitamin D promotes AVF maturation.

DETAILED DESCRIPTION:
Hemodialysis vascular access dysfunction is a major source of morbidity and cost among ESRD patients, accounting for up to 25% of all hospital stays, and 50% of all costs within the first year of initiating dialysis.The AVF provides higher blood flow rates, fewer thrombotic and infectious complications, and lower morbidity and cost compared with prosthetic grafts or central venous catheters.However,up to 50% of newly created AVF's fail to mature sufficiently for chronic hemodialysis use. Clearly, determining factors predictive of poor AVF maturation are important from both patient care and health policy perspectives and are worthy of investigation.

Vitamin D has antiproliferative, antioxidant and antiangiogenic properties. The observed association of vitamin D deficiency and increased risk of cardiovascular and peripheral vascular disease may extend to the vasculature used in the creation of an AVF.

As renal function worsens, patients with chronic kidney disease (CKD) produce less vitamin D, due to impaired renal conversion of 25-hydroxy- to 1,25-dihydroxyvitamin D by declining renal 1-alpha hydroxylase. As a result, at the time of dialysis initiation,78%-90% of ESRD patients are vitamin D deficient. Until recently, vitamin D deficiency among CKD and ESRD patients was only treated if hyperparathyroidism was present, however, more attention is now paid to nutritional vitamin D deficiency given its association with a range of comorbid conditions.Furthermore, 1,25-dihydroxyvitamin D and its analogue compounds are associated with improved survival in the CKD and ESRD populations. We believe that the observed benefits of vitamin D may improve AVF maturation among a population in which vitamin D deficiency is highly prevalent.

ELIGIBILITY:
Inclusion Criteria

* Patients with patients with end-stage renal disease (ESRD) who are suitable candidates for AVF creation (as assessed by pre-operative vein mapping) and plan to undergo AVF creation are eligible to participate
* Study subjects must agree to participate in the study and provide written informed consent
* Age: Study subjects must be > 18 years old
* Sites: Emory University affiliated hospitals (including Emory University Hospital, Emory Midtown Hospital, Grady Memorial Hospital) and Emory University affiliated outpatient dialysis units
* Informed consent requirements: All study subjects must agree to participate in the study and provide written informed consent.

Exclusion Criteria

* Age < 18 years
* Patients with a corrected serum calcium > 10.5 mg/dL within 4 weeks of study screening
* Current intake of > 2000 IU per day of Vitamin D3
* Subjects unable to provide informed consent or who plan to relocate outside of Atlanta during the study duration

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haimanot Wasse, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Mohamed I, Kamarizan MFA, Da Silva A. Medical adjuvant treatment to increase patency of arteriovenous fistulae and grafts. Cochrane Database Syst Rev. 2021 Jul 23;7(7):CD002786. doi: 10.1002/14651858.CD002786.pub4. PMID 34298589
- [Derived] Wasse H, Huang R, Long Q, Zhao Y, Singapuri S, McKinnon W, Skardasis G, Tangpricha V. Very high-dose cholecalciferol and arteriovenous fistula maturation in ESRD: a randomized, double-blind, placebo-controlled pilot study. J Vasc Access. 2014 Mar-Apr;15(2):88-94. doi: 10.5301/jva.5000187. Epub 2013 Oct 7. PMID 24101420
- [Derived] Wasse H, Huang R, Long Q, Singapuri S, Raggi P, Tangpricha V. Efficacy and safety of a short course of very-high-dose cholecalciferol in hemodialysis. Am J Clin Nutr. 2012 Feb;95(2):522-8. doi: 10.3945/ajcn.111.025502. Epub 2012 Jan 11. PMID 22237061

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 107 Assessed for Eligibility with 55 Excluded for declining to participate (12), not meeting criteria (41), and other reasons (6) leaving 52 patients randomly assigned for the study. Some individuals were counted as having more than two reasons to be excluded from the study.
Period: Overall Study
Arm/Group | Placebo | Cholecalciferol
Started | 27 | 25
Completed | 24 | 20
Not Completed | 3 | 5
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not receive vascular access type | 1 | 2
Not completed — Relocated before study completion | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cholecalciferol | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (14.9) | 49.9 (10.9) | 51.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 18 | 20 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 19 | 40
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Arteriovenous Fistulae Maturation
Description: Maturation of an AVF is the ability to stick the AVF with two large bore needles at ≥ 6 consecutive dialysis sessions, and achievement of an AVF blood flow >300 ml/min, assessed at six months following AVF creation.
Time Frame: 6 months
Measure: Number; unit: percentage of group
Arm/Group | Placebo | Cholecalciferol
Number analyzed (Participants) | 24 | 20
percentage of group | 50 | 40

2. Secondary Outcome: 25-hydroxyvitamin D and Serum Calcium
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Cholecalciferol
Number analyzed (Participants) | 24 | 20
ng/mL
  Serum 25 (OH) D | 18.4 (7.4) | 53.4 (17.7)
  Serum Calcium | 9.1 (0.6) | 8.8 (0.9)

ADVERSE EVENTS:
Arm/Group | Placebo | Cholecalciferol
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes